CLINICAL TRIAL: NCT01522612
Title: Treatment of Patients With KRAS Wild Type Advanced Colorectal Cancer (CRC) With 5-Fluorouracil (5-FU) or 5- FU Plus an Epidermal Growth Factor Receptor (EGFR) Inhibitor (Cetuximab) Based on a Comprehensive Geriatric Assessment (CGA).
Brief Title: Colorectal Cancer (CRC) Cetuximab Elderly Frail
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-40085-75083; 2011-002947-83 (EudraCT Number)
Record Dates: First submitted 2012-01-27; First posted 2012-01-31 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Colorectal Cancer Metastatic
Keywords: KRAS Wild Type; Frail Elderly; QLQ-C30; QLQ-ELD14; CGA; EGFR; Cetuximab; 5-FU
MeSH Terms: interventions — Cetuximab; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-fluorouracil/leucovorin plus cetuximab (Experimental)
  Interventions: Drug: Cetuximab; Drug: 5-fluorouracil; Drug: leucovorin
- 5-fluorouracil/leucovorin alone (Active Comparator)
  Interventions: Drug: 5-fluorouracil; Drug: leucovorin

INTERVENTIONS:
Drug: Cetuximab — 500 mg/m2 on day 1, Every 14 days Intravenously
  Other Names: Erbitux
  Arms: 5-fluorouracil/leucovorin plus cetuximab
Drug: 5-fluorouracil — Every 2 weeks, 400 mg/m2 on day 1; 2400 mg/m2 from day 1 to day 3, intravenously
  Other Names: 5-FU
Drug: leucovorin — Every 2 weeks, Racemic leucovorin 200 mg/m2 or l-leucovorin 100 mg/m2 on day 1, intravenously
  Other Names: Folinic Acid

SUMMARY:
OBJECTIVE: The principal objective of the trial is to evaluate whether the addition of cetuximab associated with 5-fluorouracil in elderly patients with KRAS wild type advanced colorectal cancer (CRC) prolongs Progression Free Survival, compared with 5-fluorouracil alone.

DETAILED DESCRIPTION:
The primary efficacy analyses will be performed on the Intention-to-treat population.

The safety analyses will be performed on the Safety population.

* Median PFS and OS in each treatment arm with its 95% CI, estimated by the Kaplan-Meier technique
* Response rates by treatment arm with their exact 95% CI
* IADL sum score, G8 sum score and social situation by treatment arm at baseline and at each timepoint of assessment
* QoL scores from the EORTC QLQ-C30 and QLQ-ELD14 modules by treatment arm at baseline and at each timepoint of assessment
* Safety data by treatment arm in the Safety population. Worst toxicity grade over all cycles according to the CTCAE criteria version 4.0 by treatment arm.
* Pharmaco-economics evaluation

Summary of proposed Phase II trial characteristics:

1. Total number of randomized patients: 150.
2. Total number of events at phase II analysis for primary endpoint: 110.
3. Total number of patients screened over the phase II: 250.
4. Total number of patients treated with cetuximab for the Phase II study: 75.
5. Maximum study duration: 19 months.

In the present study, HRQoL is an important secondary endpoint. The objective of the HRQoL data collection in this Phase II trial is to assess the impact of the addition of cetuximab on patients' HRQoL during treatment.

The hypothesis is that there will be no difference in patients' HRQoL between both treatment arms during treatment. The HRQoL domains (from the EORTC QLQ-C30 module) which are expected to be affected by treatment (to the same extent in both arms) are Global health status, Fatigue, Pain and Stool habits.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed metastatic colorectal cancer
* Measurable disease according to RECIST V1.1
* Histological local review and analysis of KRAS
* Age ≥ 80 or ≥ 70 in combination with functional restrictions defined as limitation in at least 2 of 8 IADL
* WHO performance status 0, 1 or 2
* Adequate bone marrow reserves, hepatic function & renal function
* Normal 12 lead ECG without clinically significant abnormalities
* Written informed consent before randomization according to ICH/EU GCP, and local, national and international regulations

Exclusion Criteria:

* Prior systemic chemotherapy for metastatic disease
* Previous exposure to EGFR or VEGF/VEGFR targeted therapy
* Patients may have received chemotherapy in the adjuvant or neoadjuvant setting (CRC). The treatment-free interval should be 6 months or more from the end of (neo-)adjuvant therapy
* Previous radiotherapy, either in the adjuvant setting or for the treatment of bone metastases, is allowed provided that the measurable lesions are outside the radiation fields
* Persistence of clinically relevant treatment-related toxicities from previous chemotherapy and/or radiotherapy (adjuvant or neo-adjuvant setting)
* Treatment with other investigational drugs or treatment in another clinical trial within the past four weeks before start of treatment or concomitantly with this trial
* Known alcohol or drug abuse
* Clinically significant cardiovascular disease
* Evidence of uncontrolled medical comorbidities despite adequate treatment
* Patients who have suffered a cerebrovascular accident or transient ischemic attack within the past 12 months
* History, within the past 5 years, of malignancies other than CRC
* Psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and followup schedule

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 19 months from first patient in
  Progression will be defined according to the "RECIST V1.1"

SECONDARY OUTCOMES:
Overall Survival | 19 months from first patient in
Response Rate | 19 months from first patient in
  according to the RECIST V1.1
Change in Instrumental Activities of Daily Living (IADL) score | 19 months from first patient in
Change in G8 geriatric assessment screening tool | 19 months from first patient in
Change in social situation | 19 months from first patient in
Score of Quality of Life (EORTC-QLQ C30 and QLQ-ELD14) | 14 days before randomization; 6 weeks, 14 weeks, 22 weeks and 38 weeks after randomization; 30 days after last treatment administration
Occurrence of adverse events | 19 months from first patient in
  Adverse events will be graded according to the "Common Terminology Criteria for Adverse events" CTCAE,version 4.0.
Health Economy assessments | 19 months from first patient in
Score of elderly minimal dataset comprehensive geriatric assessment (EMDCGA), as evaluated by G8 instrument | 14 days before randomization; 6 weeks, 14 weeks, 22 weeks and 38 weeks after randomization; 30 days after last treatment administration
Score of elderly minimal dataset comprehensive geriatric assessment (EMDCGA), as evaluated by Instrumental Activities of Daily Life (IADL) questionnaire | 14 days before randomization; 6 weeks, 14 weeks, 22 weeks and 38 weeks after randomization; 30 days after last treatment administration
Score of elderly minimal dataset comprehensive geriatric assessment (EMDCGA), as evaluated by social situation questionnaire | 14 days before randomization; 6 weeks, 14 weeks, 22 weeks and 38 weeks after randomization; 30 days after last treatment administration

CONTACTS AND LOCATIONS:
Overall Officials: Marc Peeters, MD, PhD, Study Chair — UNIVERSITAIR ZIEKENHUIS ANTWERPEN, Edegem, Belgium; Ulrich Wedding, MD, Study Chair — UNIVERSITAETSKLINIKUM JENA, Jena, Germany
Locations (3):
- AZ Turnhout - Campus Sint Elisabeth, Turnhout, Belgium
- Bank Of Cyprus Oncology Centre, Nicosia, Cyprus
- Hospital General Vall D'Hebron, Barcelona, Spain

REFERENCES:
- See also: Related Info — http://www.eortc.be/clinicaltrials/details.asp?protocol=40085